CLINICAL TRIAL: NCT05501808
Title: Color Stability of Two Different Resin Matrix Ceramics: Randomized Clinical Trial.
Brief Title: Color Stability of Two Different Resin Matrix Ceramics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fayoum University (Other)
Responsible Party: Principal Investigator, Alshaimaa Ahmed shabaan, associate professor in oral & maxillofacial Surgery Department, Fayoum University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: COST 315
Record Dates: First submitted 2022-08-12; First posted 2022-08-15 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2022-08

CONDITIONS: Dental Restoration
Keywords: ceramics; color; stability; resin Matrix
MeSH Terms: interventions — ENAMIC

STUDY DESIGN:
Intervention Model Description: patient with endo treated first molar
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Enamic group (Experimental): patient in this group received a restoration with enamic material
  Interventions: Procedure: enamic
- Cerasmart group (Active Comparator): patient in this group received a restoration with Cerasmart material
  Interventions: Procedure: cerasmart

INTERVENTIONS:
Procedure: cerasmart — the patient received a crown made of cerasmart ceramic
  Arms: Cerasmart group
Procedure: enamic — the patient received a crown made of enamic ceramic
  Arms: Enamic group

SUMMARY:
This is in vivo study aimed to evaluate the color stability of the newly introduced resin ceramic matrix (cerasmart )& (vita-enamic ) after a one year

DETAILED DESCRIPTION:
This is in vivo randomized clinical trial aimed to evaluate the color stability and patient satisfaction of the newly introduced resin ceramic matrix (cerasmart )& (vita-enamic ) in posterior endodontically treated teeth through one year follow-up

ELIGIBILITY:
Inclusion Criteria:

* diagnose need for restoration in endo treated posterior teeth
* good general health and oral health
* occlusal stability

Exclusion Criteria:

* smoking
* pregnancy
* use drugs that affect oral health
* Para functional habits

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 102 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
color change | 12 months
  measurement of restoration using digital spectrophotometer

SECONDARY OUTCOMES:
patient satisfaction | 12 months
  patient satisfaction is measured self questionnaire to patient consist of 5 questions with 4 answers each answer take a score from 1 to 5 where 1 is the patient is not satisfied at all and 5 is the patient is totally satisfied

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry- Fayoum University, Al Fayyum, Faiyum Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kanat-Erturk B. Color Stability of CAD/CAM Ceramics Prepared with Different Surface Finishing Procedures. J Prosthodont. 2020 Feb;29(2):166-172. doi: 10.1111/jopr.13019. Epub 2019 Jan 24. PMID 30638286
- [Background] Jorquera GJ, Atria PJ, Galan M, Feureisen J, Imbarak M, Kernitsky J, Cacciuttolo F, Hirata R, Sampaio CS. A comparison of ceramic crown color difference between different shade selection methods: Visual, digital camera, and smartphone. J Prosthet Dent. 2022 Oct;128(4):784-792. doi: 10.1016/j.prosdent.2020.07.029. Epub 2021 Mar 17. PMID 33741142
- [Derived] Mahrous AI, Salama AA, Shabaan AA, Abdou A, Radwan MM. Color stability of two different resin matrix ceramics: randomized clinical trial. BMC Oral Health. 2023 Sep 14;23(1):665. doi: 10.1186/s12903-023-03364-6. PMID 37710194